CLINICAL TRIAL: NCT03075683
Title: Internet-based Cognitive Behavioural Therapy for Insomnia in Chronic Pain: a Randomised Controlled Trial
Brief Title: Internet-based CBT for Insomnia in Chronic Pain
Acronym: IBIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/510
Record Dates: First submitted 2017-03-02; First posted 2017-03-09 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Chronic Insomnia; Chronic Pain
Keywords: Cognitive behavioural therapy; Non-pharmacological treatment; Internet mediated
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioural therapy (Experimental): Internet-based cognitive behavioural therapy for insomnia
  Interventions: Behavioral: Cognitive behavioural therapy
- Applied relaxation (Active Comparator): Internet-based applied relaxation
  Interventions: Behavioral: Applied relaxation

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — Eight sessions of internet-based CBT for insomnia comorbid with chronic pain, with active therapist support.
  Arms: Cognitive behavioural therapy
Behavioral: Applied relaxation — Eight sessions of internet-based applied relaxation for insomnia comorbid with chronic pain, with active therapist support.
  Arms: Applied relaxation

SUMMARY:
The main goal is to study the effect of therapist-guided internet-delivered cognitive behavioural therapy for insomni comorbid with chronic pain in a clinical sample.

DETAILED DESCRIPTION:
Both chronic pain and sleep disorders are prevalent and potentially very debilitating problem. The prevalence of insomnia in people with chronic pain seems to be about 50%, but figures up to 88% have been reported. Cognitive behavioral therapy for insomnia (CBT-I) has been shown to be an effective treatment for both primary insomnia and co-morbid insomnia. CBT-I is a psychotherapeutic multicomponent treatment that seeks to influence the behaviors and cognitions which perpetuates the problem. Usually, the treatment is 6-8 weeks long with one session a week, individually or in a small group setting.

Internet Mediated CBT-I has been shown to be an effective alternative to more traditional CBT. How well internet mediated CBT-I work for individuals with insomnia and co-morbid chronic pain has however not previously been investigated. The aim of the project is to study the effects of internet mediated cognitive behavioral therapy for individuals with insomnia and co chronic benign pain. The aim is to compare the effect of Internet-mediated cognitive behavioral therapy with a group that offered internet-based relaxation training. CBT-I comprises eight modules with evidence-based treatment components for insomnia (e.g. sleep restriction, stimulus control and cognitive techniques). The relaxation training comprises eight modules of applied muscular relaxation.

Hypothesis: Patients suffering from both insomnia and chronic benign pain gets significantly better treatment outcome with respect to insomnia symptoms if they receive internet-based cognitive behavioral therapy compared to those receiving internet mediated relaxation training.

Primary outcome measure: the Insomnia Severity Index (ISI), a well-used, valid and reliable self-report scale, which has been shown possible to administer via internet.

ELIGIBILITY:
Inclusion Criteria:

* Chronic insomnia Chronic benign pain No or stable pharmacological treatment for insomnia and or pain

Exclusion Criteria:

* Participation in pain management programme Pregnancy Shift work Untreated medical or psychiatric disease or disorder that could be negatively affected by insomnia treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | 8 weeks
  A well-used, valid and reliable self-report questionnaire with seven items concerning subjective symptoms and consequences of insomnia ranging from 0 to 28 points.

SECONDARY OUTCOMES:
Sleep latency | 8 weeks
  Time to fall asleep (in minutes), derived from sleep diaries.
Wake time after sleep onset | 8 weeks
  Wake time during the night (in minutes), derived from sleep diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Bothelius, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No